CLINICAL TRIAL: NCT02762773
Title: Does Avoiding Inferior Rectus Sheath Dissection Lead to Decreased Operative Blood Loss and Operating Time Without Increasing Delivery of Fetus in Primary Cesarean Delivery
Brief Title: Effect of Non-Dissection of the Inferior Rectus Sheath on Intraoperative Blood Loss
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: unable to complete recruitment
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Martin Wieczorek (Unknown)
Responsible Party: Principal Investigator, Emily Daggett, Principal Investigator, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UHCASEMC2
Record Dates: First submitted 2016-05-03; First posted 2016-05-05 (Estimated); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Acute Blood Loss Anemia; Postoperative Pain; Pregnancy
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Patients will undergo non-dissection of the inferior rectus sheath at time of primary cesarean delivery
  Interventions: Procedure: non-dissection of inferior rectus sheath
- Control (Placebo Comparator): Patients will undergo standard practice which is dissection of the superior and inferior rectus sheath at time of cesarean delivery
  Interventions: Procedure: control

INTERVENTIONS:
Procedure: non-dissection of inferior rectus sheath — Non-dissection of inferior rectus sheath
  Arms: Experimental
Procedure: control — Dissection of inferior and superior aspect of the rectus sheath
  Arms: Control

SUMMARY:
The purpose of this study is to evaluate the effect of non-dissecting the inferior rectus sheath during primary cesarean delivery on post-operative hemoglobin and post-operative pain control as measured by VAS score and opioid anesthesia use in the first 72 hours post-op.

ELIGIBILITY:
Inclusion Criteria:

* - Patients must be 18 years or older as well as willing and able to provide informed consent
* Patients undergoing a scheduled or non-scheduled, non-urgent or non-scheduled urgent (delivery within 30 minutes of decision for surgical delivery) Cesarean delivery between >35 weeks gestational age,
* Patients who are expected to receive a Pfannenstiel incision
* Patients with viable singleton intra-uterine pregnancy
* Patients with fetus in cephalic presentation

Exclusion Criteria:

* - Patients younger than 18 years,
* Patients unable or unwilling to provide informed consent,
* Patients who are illiterate,
* Patients who are non-English speaking or reading,
* Patients who are medical or nursing students at a school affiliated with University Hospital
* Multi-fetal gestations (>1 intrauterine pregnancy),
* Patients with a BMI >50 kg/m^2
* Patients with a suspected placenta accreta or placenta previa
* patients with 2 prior cesarean deliveries
* Patient undergoing emergent cesarean delivery (delivery within 10 minutes of decision for surgical delivery)
* Patients who will require a vertical skin incision, Maylard or Cherney incisions
* Patients with a history of significant pelvic adhesive disease, as determined by prior operative reports
* Patients with fetus in non-cephalic presentation
* Patients with pre-gestational or gestational diabetes mellitus
* Patients with estimated fetal weight >5000 grams
* Patients with estimated fetal weight <10% for gestational age
* Patients with who require general anesthetic
* Patients who are on chronic pain medication
* Patients with a history of drug abuse

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
post-operative hemoglobin | 24 hours
  assessment of drop in hemoglobin post-operatively compared to pre-operative values

SECONDARY OUTCOMES:
assessment of Visual Analog Scale (VAS) scores in first 72 hours | 72 hours
  assessment of VAS scores and
Assessment of total narcotic use, expressed as morphine equivalents | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Martin Wieczorek, MD, Study Director — University Hospitals Cleveland Medical Center; Melissa March, MD, Study Chair — University Hospitals Cleveland Medical Center
Locations (1):
- UH Cleveland Medical Center, Cleveland, Ohio, United States